CLINICAL TRIAL: NCT05043649
Title: A Phase 1b, Open-label, Dose-escalation Clinical Study Evaluating the Safety of Camsirubicin With Prophylactic Pegfilgrastim in the Treatment of Advanced Soft Tissue Sarcomas
Brief Title: Camsirubicin + Pegfilgrastim to Determine MTD in ASTS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of timely enrollment
Sponsor: Monopar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNPR-201-001
Record Dates: First submitted 2021-08-31; First posted 2021-09-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Advanced Soft-tissue Sarcoma
Keywords: Sarcoma; ASTS; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Camsirubicin + pegfilgrastim (Experimental): Camsirubicin phase 1b dose escalating to determine MTD
  Interventions: Drug: Camsirubicin

INTERVENTIONS:
Drug: Camsirubicin — The dose escalation of camsirubicin will start at 265 mg/m2, with dose increments of 50% until a Grade 2 non-hematologic toxicity is observed at which point subsequent dose escalations will be in increments of 25% until an MTD is identified in patients with ASTS.

SUMMARY:
This is an Interventional Study in Advanced Soft Tissue Sarcomas (ASTS). It is a Phase 1b, open-label, dose-escalation clinical study evaluating the safety of camsirubicin with prophylactic pegfilgrastim in the treatment of advanced soft tissue sarcomas. The objective of the study is to evaluate the safety of camsirubicin with prophylactic pegfilgrastim in the treatment of ASTS and determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of camsirubicin with prophylactic pegfilgrastim. The primary endpoint is the MTD (RP2D).The secondary endpoints are: safety profile of camsirubicin with prophylactic pegfilgrastim, PFS, TTP, ORR, DoR, OS and PK. As exploratory endpoint, Quality of life will be measured by using the Functional Assessment of Cancer Therapy: General (FACT-G).

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, dose-escalation clinical study evaluating the safety of camsirubicin with prophylactic pegfilgrastim in the treatment of advanced soft tissue sarcomas. Following a screening period of up to 28 days, eligible patients will receive camsirubicin through intravenous (IV) infusion (8 mL/min rate) once every 21 days, starting on Day 1 of a 21-day cycle for 6 cycles. Dose will be based on the patient's body surface area (BSA). Patients who demonstrate clinical benefit (defined as stable disease or better) at the completion of 6 cycles will be allowed to continue to receive camsirubicin until disease progression or unacceptable toxicity. All patients receiving camsirubicin will also receive 6 mg of prophylactic pegfilgrastim approximately 24-96 hours after each camsirubicin infusion to prevent neutropenia. The dose escalation will start at 265 mg/m2, with dose increments for subsequent dose groups of 50% until a drug-related Grade 2 non-hematologic toxicity is observed, at which point subsequent dose escalations will be in increments of 25% until an MTD is identified.

At each successive dose level, cohorts of 3 new patients will be entered if no dose-limiting toxicity (DLT) is observed (3+3 design) within 21 days of initial dose. If a patient treated at any dose level experiences a DLT, a total of up to 6 patients will be treated at that dose level. Once two patients at any dose level experience a DLT, no additional patients will be treated at that level. The MTD is defined as the highest dose level below the dose level at which 2 or more patients experience a DLT during the first 21 days from Cycle 1 Day 1. This will be the RP2D unless safety concerns suggest a lower dose. Patients in each new cohort at all dose levels (i.e., all patients receiving their initial dose of camsirubicin at the designated dose level) will successfully complete one cycle of treatment prior to beginning treatment of the new cohort of patients at the next higher dose level.

The RP2D dose may be expanded by 6 patients to obtain additional PK and safety data at this dose. Patients will be followed for adverse events of special interest (AESI), which include the incidence of congestive heart failure (CHF) and left ventricular ejection fraction (LVEF) dysfunction. Patients will be followed for 1 year post last dose and AESI assessed every 3 months. Assessments will include LVEF assessment by echocardiogram or multi-gated radionuclide angiography (MUGA) scan and measurement of Troponin-I. LVEF assessments should be collected even if the patient will go on to other anticancer therapies during the 1-year post last dose long-term follow-up period. If cardiac toxicity is suspected, an echocardiogram should be performed sooner if a patient develops signs and symptoms of congestive heart failure (e.g., shortness of breath during mild exertion or when lying down, feel very tired, cough (especially at night), swelling of the feet and/or ankles).

Patients with serious adverse events (SAEs) or AESI assessed by the investigator during the 1-year follow-up period as related to study medications will be followed until the AE completely resolves or is assessed as chronic. Unresolved SAE or AESI at the end of the 1-year long-term follow-up period will be followed for status for up to 2 years at approximately 3-month intervals.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for inclusion in this study:

1. The participant must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g., blood count, imaging tests) and obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age ≥18 years.
3. Only locally confirmed histological diagnosis of advanced unresectable or metastatic malignant soft tissue sarcoma (including leiomyosarcoma, dedifferentiated liposarcoma, myxoid liposarcoma, pleomorphic liposarcoma, undifferentiated pleomorphic sarcoma, malignant peripheral nerve sheath tumor, high-grade sarcoma [not otherwise specified], or synovial sarcoma) not amenable to curative treatment with surgery or radiotherapy.
4. Presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
5. Performance status 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
6. The participant has not received any previous treatment with anthracyclines (not even in adjuvant therapy).
7. The participant has not had any prior systemic cytotoxic therapies for advanced/metastatic sarcoma and is considered an appropriate candidate for anthracycline therapy. All previous anticancer treatments must be completed ≥28 days prior to first dose of study drug.
8. Laboratory tests must be as follows and may be repeated once at the discretion of the investigator:

   1. Absolute neutrophil count (ANC) ≥1,500/mm³
   2. Platelet count ≥100,000/mm³
   3. Hemoglobin >9 g/dL
   4. Bilirubin <1.5 times upper limit of normal (ULN); except subjects with Gilbert Syndrome who must have a total bilirubin level <3.0 x ULN
   5. Prothrombin time (PT) (seconds) or international normalized ratio (INR) ≤1.5 x ULN
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN or, in patients with documented hepatic metastasis, ≤5 x ULN
   7. Serum creatinine ≤1.5 mg/dL or estimated creatinine clearance ≥60 mL/min (Cockroft and Gault)
9. Left ventricular ejection fraction (LVEF) ≥50% assessed within 28 days prior to enrollment.
10. Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment. A female is eligible to enter and participate in the study if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had a hysterectomy, a bilateral oophorectomy (ovariectomy), a bilateral tubal ligation, or is postmenopausal with a minimum of 1 year without menses.
11. Both males and females must agree to use highly effective contraceptive precautions if conception is possible during the dosing period and up to 3 months following the last dose of study drug.
12. Female patients who are lactating must agree to discontinue nursing prior to the first dose of study drug and must refrain from nursing throughout the treatment period and for 3 months following the last dose of study drug.
13. The participant has, in the opinion of the investigator, a life expectancy of at least 3 months.

Exclusion Criteria:

Patients must not meet any of the exclusion criteria to be eligible for study participation.

1. Current evidence/diagnosis of alveolar soft part sarcoma, extraskeletal myxoid chondrosarcoma, rhabdomyosarcoma, osteosarcoma, gastrointestinal stromal tumor (GIST), dermatofibrosarcoma (unless transformed to fibrosarcoma), Ewing's sarcoma, Kaposi's sarcoma, mixed mesodermal tumor, or clear cell sarcomas.
2. Patients who cannot tolerate pegfilgrastim.
3. Known active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of enrollment. Participants with a history of a CNS metastasis previously treated with curative intent (e.g., stereotactic radiation or surgery) that have not progressed on follow-up imaging, have been asymptomatic for at least 60 days prior to first dose, and are not receiving systemic corticosteroids and or/anticonvulsants are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before enrollment to rule out brain metastasis.
4. Prior treatment with doxorubicin, epirubicin, idarubicin, and/or other anthracyclines or anthracenediones (including adjuvant therapy).
5. Prior radiotherapy of the mediastinal/pericardial area or whole pelvis radiation. Other thoracic radiotherapy is permitted.
6. The participant has symptomatic congestive heart failure (CHF), left ventricular ejection fraction dysfunction (LVEF <50%), severe myocardial insufficiency, cardiac arrhythmia (uncontrolled, clinically significant), or cardiomyopathy.
7. The participant has unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction within 6 months of enrollment.
8. The participant has a QT interval calculated using Fridericia's correction (QTcF) of >450 milliseconds (msec) for males and >470 msec for females on screening electrocardiogram (ECG).
9. Females who are pregnant or breastfeeding.
10. Known allergy to any of the treatment components including a history of allergic reactions attributed to compounds of chemical or biological composition similar to doxorubicin and camsirubicin, including intravenous (IV) lactose, or pegfilgrastim.
11. The participant has a known, uncontrolled active fungal, uncontrolled bacterial, or uncontrolled viral infection including human immunodeficiency virus (HIV) or viral hepatitis (B or C).
12. Any malignancy other than soft tissue sarcoma within the last 5 years prior to screening, with the exception of:

    1. Cervical carcinoma in situ or
    2. Basal cell carcinoma or
    3. Superficial bladder tumors that have been successfully and curatively treated with no evidence of recurrent or residual disease.
13. Unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, confound the assessment of camsirubicin's effect, jeopardize the safety of a patient and/or their compliance with the protocol.
14. Currently receiving any investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
To determine Maximum Tolerated Dose (MTD) | 3 weeks after first injection
  Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0) will be collected for all treated subjects at each dose level of camsirubicin to identify dose limiting toxicities (DLTs). At each successive dose level, cohorts of 3 new patients will be entered if no dose limiting toxicity (DLT) is observed (3+3 design) within 21 days of initial dose. If a patient treated at any dose level experiences a DLT, a total of up to 6 patients will be treated at that dose level. Once two patients at any dose level experience a DLT, no additional patients will be treated at that level. The MTD will be defined as the highest dose level below the dose level at which 2 or more patients experience a DLT during the first 21 days from Cycle 1 Day 1.
Recommended Phase 2 Dose (RP2D) Camsirubicin HCl for Injection | Up to 1 year after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the safety expansion cohort, based on safety, tolerability, efficacy, PK, and MTD data collected during the dose escalation portion of the study.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | Up to 1 year after the first dose
  Safety profile of camsirubicin with prophylactic pegfilgrastim, through assessment of adverse event (AE) type, incidence, severity, time of appearance, and related causes (detected by physical explorations and laboratory tests). Adverse events will be graded and tabulated using NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Holli Carlson, Study Director — Monopar Therapeutics Inc.
Locations (2):
- United States (2):
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Washington Medicine Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No